CLINICAL TRIAL: NCT02050776
Title: The Role of Cell Therapy in Modifying the Course of Limb Girdle Muscular Dystrophy- A Longitudinal 5-year Study
Brief Title: Stem Cell Therapy in Limb Girdle Muscular Dystrophy
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Sponsor: Neurogen Brain and Spine Institute (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NGBSI-07
Record Dates: First submitted 2014-01-29; First posted 2014-01-31 (Estimated); Last update posted 2018-10-25 (Actual); Status verified 2018-10

CONDITIONS: Limb Girdle Muscular Dystrophy
MeSH Terms: conditions — Muscular Dystrophies, Limb-Girdle

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Stem Cells (Experimental): autologous bone marrow mononuclear cell transplantation
  Interventions: Biological: Autologous bone marrow mononuclear cell transplantation

INTERVENTIONS:
Biological: Autologous bone marrow mononuclear cell transplantation — bone marrow derived mononuclear cells are administered intrathecally and intramuscularly in limb girdle muscular dystrophy patients

SUMMARY:
The purpose of this study was to study the effect of stem cell therapy on the course of the disease in patients with Limb Girdle Muscular Dystrophy.

ELIGIBILITY:
Inclusion Criteria:

* males and females
* age group of 15 years and above
* limb girdle muscular dystrophy diagnosed on the basis of clinical presentation
* Electromyographic and Nerve Conduction velocity findings

Exclusion Criteria:

* presence of respiratory distress
* presence of acute infections such as Human Immunodeficient Virus/Hepatitis B Virus/Hepatitis C Virus
* malignancies
* acute medical conditions such as respiratory infection, fever, hemoglobin less than 8, bleeding tendency, bone marrow disorder, left ventricular ejection fraction < 30%
* pregnancy or breastfeeding

Ages: 15 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 0 (Actual)
Dates: Start 2008-12; Primary Completion 2013-03 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
Functional Independence Measure | 6 months

SECONDARY OUTCOMES:
Manual Muscle Testing | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Alok K Sharma, M.S., M.Ch, Principal Investigator — Neurogen Brain and Spine Institute
Locations (1):
- Neurogen brain and spine institute, Mumbai, Maharashtra, India

REFERENCES:
- [Background] Sharma A, Sane H, Badhe P, Gokulchandran N, Kulkarni P, Lohiya M, Biju H, Jacob VC. A clinical study shows safety and efficacy of autologous bone marrow mononuclear cell therapy to improve quality of life in muscular dystrophy patients. Cell Transplant. 2013;22 Suppl 1:S127-38. doi: 10.3727/096368913X672136. Epub 2013 Sep 10. PMID 24070109